CLINICAL TRIAL: NCT03749525
Title: Effect of Shenfu Injection on Arterial Vascular Reactivity in Patients With Septic Shock
Brief Title: Shenfu Injection Improves Arterial Vascular Reactivity
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jianfeng Xie (Other)
Responsible Party: Sponsor-Investigator, Jianfeng Xie, physician, sponsor-investigator,clinical professor, Southeast University, China
Organization: Southeast University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: shenfu injection
Record Dates: First submitted 2018-07-09; First posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Septic Shock; Shenfu; Vascular Reactivity
MeSH Terms: conditions — Shock, Septic | interventions — Shen-Fu

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo group (Placebo Comparator): 5% GS solution
  Interventions: Drug: shenfu injection
- control group (Active Comparator): shenfu injection
  Interventions: Drug: shenfu injection

INTERVENTIONS:
Drug: shenfu injection — we hypothesis that shenfu injection could improve patients' arterial vascular reactivity with septic shock
  Other Names: 5% GS solution

SUMMARY:
Septic shock is a common and critical illness in ICU.The vascular dysfunction of septic shock is manifested by vasospasm and decreased arterial vascular reactivity . Current studies have shown that the main mechanisms of vasospasm and decreased arterial vascular reactivity include increased vasospasm and down-regulation of receptor sensitivity , and eventually cause a decrease in vascular smooth muscle contractility.A large number of vasodilators are released during septic shock, in which inducible nitric oxide synthase (iNOS) and prostacyclin (PGI2) are important vasodilators leading to septic shock vasospasm.At present, vasoactive drugs are widely used in clinically to improve vascular tone and are important means of circulation support. However, when the infection is heavier, the reactivity of the blood vessels to the vasoactive drugs is lowered, and it is difficult for the large doses of the vasoactive drugs to maintain the circulation stability. At this time, the use of vasoactive drugs alone does not benefit patients with septic shock and may require the combination of other drugs.From the perspective of Chinese medicine, shock is a disease of yang. Shenfu injection has the effect of rejuvenating the yang and replenishing the qi. This trial was designed to give patients with septic shock the use of Shenfu injection to determine the specific effects of Shenfu injection on vascular reactivity in patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed as septic shock according to 2016 SSC Guidelines;
2. The dose of norepinephrine required to maintain MAP>65mmHg ≥0.5μg/kg.min;
3. SVRI <800 dyns/cm5.m2;
4. CI>2.5L/min/m2;
5. The patient or the patient's family signed the informed consent form for this trial.

Exclusion Criteria:

1. septic shock occurs more than 24 hours;
2. Age > 85 years old or <18 years old;
3. pregnant or lactating women;
4. There are shock patients caused by other causes such as cardiogenicity and neurogenicity;
5. The terminal state of malignant tumor end-stage disease or the patient who is expected to die within 24 hours.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Han
Enrollment: 26 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
The change of peripheral vascular resistance | day 0(before shenfu injection is used), day 3 (after shenfu injection is used for 72 hours)
  Peripheral vascular resistance will be measured by PiCCO or Swan-Ganz and the change between day 0 and day 3

SECONDARY OUTCOMES:
Diastolic blood pressure | day 1, day 2, day 3
  We will measure blood pressure every hour and diastolic blood pressure will be recorded per hour.
Dosage of vasoactive drugs | day 1, day 2,day 3
  dosages of noradrenaline, adrenaline or any other kinds of vasoactive drugs
  4/5000 dosages of adrenaline and norepinephrine

CONTACTS AND LOCATIONS:
Overall Officials: haibo qin, professor, Study Chair — southeast university zhongda hospitial

IPD SHARING:
Plan to Share IPD: Undecided